CLINICAL TRIAL: NCT07050277
Title: Post-Operative Urinary Retention on Revision Knee Arthroplasty: the Role of Intrathecal Morphine
Acronym: POURRKA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Hermann dos Santos Fernandes, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MSH REB # 0065
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Arthroplasties, Knee Replacement; Nerve Block; Urinary Retention Postoperative; Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrathecal Morphine (Active Comparator): Adductor canal block; IPACK block; Spinal anesthesia: Isobaric Bupivacaine 0.5% 2.5 mL + Fentanyl 15 mcg + Morphine 100 mcg
  Interventions: Drug: Intrathecal Morphine
- No Intrathecal Morphine (Experimental): Adductor canal block; IPACK block; Spinal anesthesia: Isobaric Bupivacaine 0.5% 2.5 mL + Fentanyl 15 mcg
  Interventions: Drug: No Intrathecal Morphine

INTERVENTIONS:
Drug: Intrathecal Morphine — Intrathecal morphine
  Arms: Intrathecal Morphine
Drug: No Intrathecal Morphine — No Intrathecal Morphine
  Arms: No Intrathecal Morphine

SUMMARY:
Revision total knee arthroplasty (rTKA) is a frequently performed procedure. Adequate pain management is an important feature, especially for fast-track and Enhanced Recovery After Surgery (ERAS) programs. The multimodal approach, including single shot or continuous nerve blocks with catheters and spinal or epidural morphine, is a stablished strategy. Although the administration of intrathecal morphine (IM) has been shown to significantly reduce pain scores, it is not free of adverse effects. Postoperative urinary retention (POUR) is possible and might increase the risk of periprosthetic infection. The purpose of this study is to compare patients undergoing rTKAS under spinal anesthesia with IM to patients undergoing the same procedure, under the same anesthetic technique, but with no IM, for POUR and postoperative pain related outcomes. All patients will have single shot and continuous adductor canal block (CACB) and single shot IPACK (interspace between the popliteal artery and the posterior knee capsule) block. The hypothesis is that postoperative pain control is comparable between the groups, with lower incidence of POUR in patients with no IM given.

DETAILED DESCRIPTION:
Introduction Total knee arthroplasties (TKA) are among the most performed surgeries worldwide(1). In Canada, between 2020 and 2021, 55,285 TKAs were performed, with 4179 (7.56%) being revision total knee arthroplasties (rTKA). The main reasons for rTKAs are infection (35.6%), aseptic loosening (18.0%) and instability (3.6%)(2). Most TKA are done under a neuraxial anesthetic technique alongside a multimodal approach to postoperative pain management. The approach to postoperative pain management comprises combining intrathecal opioids like morphine, fentanyl; IPACK (interspace between the popliteal artery and the posterior knee capsule) block; adductor canal block (ACB), single shot or continuous with catheters; local infiltration analgesia (LIA) and systemic administration of paracetamol and non-steroid anti-inflammatory drugs (NSAIDs). Oral and intravenous (IV) opioids are usually reserved as rescue medications(3).

In many types of surgeries (lower limbs and abdominal surgeries), intrathecal morphine (IM) administration has been shown to significantly reduce pain scores and postoperative opioid requirements within the first 24 hours. However, its administration has potential side effects, which includes respiratory depression, pruritus, nausea, vomiting and postoperative urinary retention (POUR)(4-7). POUR may require bladder catheterization and can result in delayed hospital discharge and poor patient satisfaction. Ultimately, the need for bladder catheterization increases the risk of periprosthetic infection in hip and knee arthroplasties surgeries(8, 9).

Among primary TKA surgery, there is fair amount of evidence demonstrating equivalence of IM to femoral nerve block or ACB for postoperative analgesia, but at the cost of side effects when IM is used(10, 11). Therefore, for primary TKA surgery, when the proper peripheral nerve blocks are performed, IM is often not used.

A limitation of most of the existing literature focusing on postoperative analgesia in TKA is the exclusion of rTKA surgeries. Consequently, there are very few studies to guide analgesic management specific to rTKA. One study demonstrates that, when a multimodal protocol including continuous ACB (CACB) was performed, patients who underwent rTKA experienced a similar postoperative analgesic course as primary TKA patients(12). Regardless the benefits of peripheral nerve blocks and the potential side effects of IM, the latter is still commonly used for rTKA perioperative management. To the best of our knowledge, there is no prospective study assessing the real analgesic role and potential side effects of IM in addition to peripheral nerve blocks in rTKAs.

Significance Revision TKAs are on a rise following primary TKA. It is a more costly procedure than primary TKA and tends to be more painful. In our institution (Mount Sinai Hospital - Sinai Health System - Toronto, Ontario, Canada), most rTKAs are done under neuraxial anesthesia with IM to achieve optimal pain control. Peripheral nerve blocks (single shot and CACB and IPACK block) are done depending on the presence or absence of contra-indications (anatomy abnormalities, infection on block site). The usage of IM has been shown to be a risk factor for POUR(4, 6), which may require bladder catheterization for its management. This increases the risk for urinary tract infections and subsequently periprosthetic joint infection(8, 9). Despite of the potential side effects, IM is still fairly used for postoperative management in rTKA surgeries.

Given the current literature on the benefits of peripheral nerve blocks for postoperative pain control in primary TKAs and its equivalence to IM for postoperative pain control outcomes with lower incidence of POUR, in addition to the lack of specific evidence comparing peripheral nerve blocks and IM in rTKA, an interesting study subject is noticed. As rTKA surgery is on a rise for the future, there is significant importance in investigations on interventions which may improve recovery and decrease complications.

Objectives The objective of this study is to evaluate the effectiveness of spinal anesthesia with no IM associated with single shot ACB and IPACK block, and CACB in comparison to spinal anesthesia with IM in association with single shot ACB and IPACK block, and CACB for pain management in patients undergoing rTKA due to non-infection causes, for POUR and pain control outcomes.

Hypothesis Postoperative pain control is similar in patients undergoing non-infected rTKA performed under spinal anesthesia with IM in addition to single shot ACB and IPACK block, and CACB, when compared with patients having the same anesthesia technique with the exception of the IM, however with lower incidence of POUR when IM is not given.

Methods Study type Prospective randomized controlled trial, blinded for patient and evaluator (data collector), in patients undergoing rTKA at Mount Sinai Hospital, Sinai Health System, Toronto, ON, Canada. Recruitment of subjects will start after Research Ethics Board approval. Patients will be assessed for their eligibility to participate in the study. Clear and concise information about the study and interventions to be carried out will be given to study participants after which a signed written informed consent will be obtained.

Perioperative management and interventions Subjects booked for rTKA will be recruited during pre-anesthesia consultation in Pre-Admission Unit. The study proposal will be presented and explained to the patients on that moment. The study consent form with the study information will be given to them. They will have ample time between the pre anesthesia assessment and the surgery, to review and provide informed consent for the study. Signed informed consent will be obtained on the morning of the surgery once the patients come into the hospital.

The research participants will be randomized to one of the two groups using a computer-generated random numbers table. Randomization will be done at the start of the study and all numbers will be allocated to one of the two study groups:

1. Interventional group: no IM;
2. Control group: IM. Once the numbers are generated, the method to allocate participants to the respective study intervention will be sequentially numbered opaque sealed envelopes.

Every patient will receive a study number following the order of their entrance on the study. The researcher who collects the data and the anesthesiologist involved in patient care will be blinded to which group each patient is randomized to. A different research team member, who is not involved in patient care or in data collection, will be responsible to check the patient allocation (according to the randomization) and prepare the spinal anesthesia solution (with or without IM). All patients will receive the same perioperative management with the exception of the IM, depending on their group.

After the patients are admitted for their surgery, they will initially be brought to a dedicated block room area where a safety checklist will be performed by the block room team and patients will receive preoperative analgesic medication (PO Celecoxib 100-200 mg and Acetaminophen 1 g). Standard Canadian Anesthesia Society monitoring will be provided. Intravenous (IV) line will be inserted. Mild sedation with Midazolam 0.5 - 2 mg and Fentanyl 25-100 mcg might be administered for anxiolysis and analgesia. After proper cleaning of the ipsilateral thigh, with a sterile technique and ultrasound guidance (Sonosite Edge II ultrasound machine), an ACB (injection of 15-20 mL of Ropivacaine 0.5% with epinephrine 1:200,000) and an IPACK block (injection of 10-15 mL of Ropivacaine 0.25% with epinephrine 1:200,000) will be performed. These pre-operative nerve blocks are part of the standard of practice for perioperative management of TKAs, at Mount Sinai Hospital. Total local anesthetic doses will be pre-emptively calculated to avoid a total Ropivacaine dose of > 3 mg/kg. After the peripheral nerve blocks, all patients will receive standard spinal anesthesia (Isobaric Bupivacaine 0.5% 2.5 mL + Fentanyl 15 mcg). Depending on the group they are randomized to, they will have Morphine 100 mcg added to the spinal solution, or not. The use or absence of intrathecal Morphine are neither part of the standard of practice for perioperative management of TKAs, at Mount Sinai Hospital. The use of this agent is variable and dependable on attending anesthesiologist's preferences, impossibility of performing the specific nerve blocks or inserting the adductor canal catheter, or if patient have specific contra-indications for the neuraxial agents of for the nerve blocks. After the spinal anesthesia is performed and tested as effective, patients will be brought to the operation room. During surgery, each patient will receive IV Cefazolin 2-3 g (depending on their weight), Tranexamic acid 20 mg/kg, Dexamethasone 0.1 mg/kg, and Ondansetron 4 mg. They will be kept sedated with an IV weight-based Propofol infusion (dose range: 50-150 mg/kg/h, as needed for patient's comfort). At the end of the procedure the surgeons will infiltrate the surgical site with a solution of 200 mg Ropivacaine 0.2% and epinephrine 1:200,000.

After surgery, the patient will be taken to the Post Anesthesia Care Unit. At this moment, an Arrow® or Pajunk® catheter trough the needle CACB catheter will be inserted using a Sonosite Edge II or Sonosite X-Porte ultrasound machine. Catheters will be inserted by a staff anesthesiologist from the Regional Anesthesia Team or by a Regional Anesthesia Fellow under the regional anesthesia staff supervision accordingly with the ISAFE technique (Inter-fascial space between SArtorius and FEmoral artery)(13). During catheter insertion, 10-20 mL dextrose 5% with epinephrine 1:200,000 solution will be used for hydro dissection, intravascular injection verification, solution spread and catheter function testing. During the procedure, patient will be monitored for any heart rate change to rule out intravascular catheter placement. The catheter will be well secured with adhesive fixation device to avoid displacement. Following catheter placement, the catheter will be aspirated to check for blood to ensure there is no intravascular placement and will be aspirated prior to any injection. The peripheral nerve catheter will be connected to a Baxter elastomeric pump containing a solution of Ropivacaine 0.2%. Infusion rate will be of 5 mL/h and will be kept for a total of 48-60 hours. The patient will be monitored in the post anesthesia unit and then discharged to the ward in accordance with standard post anesthesia care unit guidelines. The adductor canal catheter will infuse for 48-60 hours. The patients will be followed up for 48 hours, counting from the spinal anesthesia injection time. The use of adductor canal catheter for CACB is part of the standard of practice for perioperative management of TKAs, at Mount Sinai Hospital.

The patient will be discharged to home after achieving the discharge criteria (being medically cleared by the physician, passing physiotherapy functional assessment, pain well controlled on oral pain medication, tolerating an oral diet without nausea or vomiting, and voiding independently). If the discharge occurs within less than 48 hours after the spinal anesthesia is performed, the patients will go home with the CACB catheter in place, connected to the elastomeric pump, with the same infusion rate, and will remove the catheter and dispose the devices when the infusion completes 48-60 hours. Prior to going home, patients will receive education and written information (educational pamphlet) regarding monitoring for local anesthetic systemic toxicity (LAST) symptoms, possible CABC associated complications including potential transient muscle weakness, and instructions on how to remove the catheter after 48-60 hours. This pamphlet will contain contact information for Acute Pain Service, in case of any events, adverse effects or questions the patients may have about the peripheral nerve catheter. And patients will be followed up for the study by a phone assessment. If patients stay in hospital for more than 48 hours after the spinal anesthesia was performed, the assessments will be done in-person and the CACB catheter will be removed when the infusion reaches 48-60 hours. While in the hospital, patients will have their postoperative analgesic prescription as the standard: Acetaminophen 650-1000 mg QID, Celecoxib 100-200 mg BID, Hydromorphone 1-2 mg PRN Q2Hs; Hydromorphone 0.2-0.8 mg IV PRN Q1Hs. When at home, their prescription will be: Acetaminophen 650-1000 mg QID, Celecoxib 100-200 mg BID, Hydromorphone 1-2 mg PRN Q4Hs.

Sample size The sample size is calculated based on a previous literature that demonstrates that IM can be associated POUR in 25-36% of cases(6). Considering an incidence of 30% of POUR in patients receiving IM and no POUR in patients with no IM given, for an alpha=0.05 and power of 80%, 21 subjects in each group would be needed for this study. Anticipating possible dropouts, 25 patients per group will be recruited for this study, with a total of 50 patients.

Study data analysis Normal distributed variables values will be presented and analyzed as mean values ± standard deviation. Non-normal distributed variables values will be presented and analyzed as median and minimum and maximum values. Qualitative variables will be presented as frequency of occurrence. Statistical test to be performed will be t-Student, Kruskal-Wallis and Chi-square. Statistical software will be used for analysis: SPSS 13.0 for Windows (SPSS Inc, Chicago, IL, USA) and GraphPad Prism Version 4.00 for Windows (GraphPad Software, San Diego, CA, USA).

ELIGIBILITY:
Inclusion Criteria:

* Non pregnant patients undergoing unilateral non infected rTKA surgery;
* Older than 21 years of age, with American Society of Anesthesiologists (ASA) physical status I-III;
* With no alcohol or drug dependency history;
* With sufficient understanding and co-operation about the usage of a perineural catheter for pain management; body mass index (BMI) under 45;
* With no allergy to medications used in the study protocol (bupivacaine, lidocaine, ropivacaine, midazolam, propofol, ketamine, morphine, hydromorphone, fentanyl, acetaminophen, celecoxib, ondansetron, dexamethasone, tranexamic acid);
* No current or recent use of opioids (within the last 2 weeks) in an average oral morphine equivalent (OME) of 20 mg/day or higher;
* With no contra-indications for neuraxial anesthesia, IPACK block, ACB and adductor canal catheter insertion;
* Who speak and understand the English language;
* Who agrees to participate on this study through the signature of the consent form.

Exclusion Criteria:

* Patients will be excluded of the study if they have a failed spinal anesthesia and needs for a conversion to general anesthesia;
* If peripheral nerve blocks are not possible to be performed due to technical difficulties;
* If during patient's care a deviation of the protocol occurs;
* If CACB catheter has issues on its function, disconnects or exteriorizes within the first 48 hours of infusion;
* Or if patient decides to withdraw from the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative urinary retention | First 48 hours after spinal anesthesia
  need of bladder catheterization at any moment

SECONDARY OUTCOMES:
Quality of Recovery | 24 and 48 hours after spinal anesthesia
  Quality of Recovery - 15 (QoR-15) scores: from 0 to 150. Higher scores mean better outcomes.
Pain at rest | 24 and 48 hours after spinal anesthesia
  Pain intensity at rest: pain intensity when patient is not moving the knee, through numerical rating scale (NRS) for pain (0 = no pain at all; 10 = worst pain)
Pain at movement | 24 and 48 hours after spinal anesthesia
  Pain intensity at movement: pain intensity when patient moves from sitting to standing position, through numerical rating scale (NRS) for pain (0 = no pain at all; 10 = worst pain)
Opioid consumption | 24 and 48 hours after spinal anesthesia
  Opioid usage in oral morphine equivalent (OME);

CONTACTS AND LOCATIONS:
Overall Officials: Hermann dos Santos Fernandes, MD, PhD, Principal Investigator — Department of Anesthesia and Pain Management, Mount Sinai Hospital Assistant
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
After finalization of the study, IPD can be shared, in a anonymized manner, with other colleagues, by request.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Lavand'homme PM, Kehlet H, Rawal N, Joshi GP; PROSPECT Working Group of the European Society of Regional Anaesthesia and Pain Therapy (ESRA). Pain management after total knee arthroplasty: PROcedure SPEcific Postoperative Pain ManagemenT recommendations. Eur J Anaesthesiol. 2022 Sep 1;39(9):743-757. doi: 10.1097/EJA.0000000000001691. Epub 2022 Jul 20. PMID 35852550
- [Background] Dana E, Ben-Zur O, Dichtwald S, Feigin G, Brin N, Markushevich M, Fredman B, Brin YS. Postoperative urinary retention following hip or knee arthroplasty under spinal anaesthesia with intrathecal morphine: a retrospective cohort study. Singapore Med J. 2025 Sep 1;66(9):481-485. doi: 10.4103/singaporemedj.SMJ-2022-108. Epub 2023 Jun 13. PMID 37338499
- [Background] Scholten R, Kremers K, van de Groes SAW, Somford DM, Koeter S. Incidence and Risk Factors of Postoperative Urinary Retention and Bladder Catheterization in Patients Undergoing Fast-Track Total Joint Arthroplasty: A Prospective Observational Study on 371 Patients. J Arthroplasty. 2018 May;33(5):1546-1551. doi: 10.1016/j.arth.2017.12.001. Epub 2017 Dec 13. PMID 29306574
- [Background] Staikou C, Paraskeva A. The effects of intrathecal and systemic adjuvants on subarachnoid block. Minerva Anestesiol. 2014 Jan;80(1):96-112. Epub 2013 Jul 9. PMID 23839318
- [Background] Tomaszewski D, Balkota M, Truszczynski A, Machowicz A. Intrathecal morphine increases the incidence of urinary retention in orthopaedic patients under spinal anaesthesia. Anaesthesiol Intensive Ther. 2014 Jan-Mar;46(1):29-33. doi: 10.5603/AIT.2014.0006. PMID 24643924
- [Background] Cha YH, Lee YK, Won SH, Park JW, Ha YC, Koo KH. Urinary retention after total joint arthroplasty of hip and knee: Systematic review. J Orthop Surg (Hong Kong). 2020 Jan-Apr;28(1):2309499020905134. doi: 10.1177/2309499020905134. PMID 32114894
- [Background] Garbarino LJ, Gold PA, Anis HK, Sodhi N, Danoff JR, Boraiah S, Rasquinha VJ, Mont MA. Does Intermittent Catheterization Compared to Indwelling Catheterization Decrease the Risk of Periprosthetic Joint Infection Following Total Knee Arthroplasty? J Arthroplasty. 2020 Jun;35(6S):S308-S312. doi: 10.1016/j.arth.2020.02.055. Epub 2020 Feb 28. PMID 32192833
- [Background] Janiak M, Kowalczyk R, Gorniewski G, Olczyk-Miiller K, Kowalski M, Nowakowski P, Trzebicki J. Efficacy and Side Effect Profile of Intrathecal Morphine versus Distal Femoral Triangle Nerve Block for Analgesia following Total Knee Arthroplasty: A Randomized Trial. J Clin Med. 2022 Nov 25;11(23):6945. doi: 10.3390/jcm11236945. PMID 36498519
- [Background] Li XM, Huang CM, Zhong CF. Intrathecal morphine verse femoral nerve block for pain control in total knee arthroplasty: A meta-analysis from randomized control trials. Int J Surg. 2016 Aug;32:89-98. doi: 10.1016/j.ijsu.2016.06.043. Epub 2016 Jul 6. PMID 27370542
- [Background] Grant AE, Schwenk ES, Torjman MC, Hillesheim R, Chen AF. Postoperative Analgesia in Patients Undergoing Primary or Revision Knee Arthroplasty with Adductor Canal Block. Anesth Pain Med. 2017 Apr 17;7(3):e46695. doi: 10.5812/aapm.46695. eCollection 2017 Jun. PMID 28824869
- [Background] Dos Santos Fernandes H, Siddiqui N, Peacock S, Vidal E, Wolfstadt J, Gleicher Y. Inter-fascial space between SArtorius muscle and FEmoral artery (ISAFE): A suggested approach for Adductor Canal catheter placement. J Clin Anesth. 2022 Feb;76:110571. doi: 10.1016/j.jclinane.2021.110571. Epub 2021 Nov 8. No abstract available. PMID 34763273